CLINICAL TRIAL: NCT00086567
Title: A Multi-Institutional Study of Proteomic Evaluation of Epithelial Ovarian Cancer, Primary Peritoneal Cancer, and Fallopian Tube Cancer Patients in First Clinical Remission: Development of a Protein Fingerprint Profile of Relapse
Brief Title: Predictors of Relapse of Ovarian, Peritoneal, and Fallopian Tube Cancers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040232; 04-C-0232; NCT00119353 (obsolete NCT alias)
Record Dates: First submitted 2004-07-02; First posted 2004-07-05 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-07-30

CONDITIONS: Fallopian Tube Cancer; Peritoneal Neoplasms; Epithelial Ovarian Cancer
Keywords: Blood; Testing; Gynecologic; Urine; CA125; Natural History; Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Peritoneal Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Patients in first remission from treatment of FIGO stage III/IV primary peritoneal, fallopian tube, or epithelial ovarian carcinoma

SUMMARY:
This study will develop a blood test that can be used to predict a relapse of ovarian, peritoneal, or fallopian tube cancer. The type of testing is called proteomics, or the study of proteins in living cells. The test will identify certain proteins that might represent a pattern, or "fingerprint," indicating increased risk of disease relapse.

Women with Stage III or IV epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer that is in remission may be eligible for this study. Candidates are screened with a medical history and physical examination, blood tests, review of pathology report from surgery, and computed tomography (CT) or magnetic resonance imaging (MRI) scans of the abdomen and pelvis (and chest if the cancer spread to the chest).

Participants have a clinic visit every 3 months for a physical examination (including a pelvic examination), blood draw for routine and research tests, and review of how they have been feeling. Every 6 months they have CT scans of the abdomen, pelvis, and possibly the chest. When a patient has been in remission for 4 years, blood draws are done every 6 months and CT scans are done yearly. Patients whose cancer returns (based on a CA-125 blood test, CT scans, or physical examination) end their participation in the study. Patients with an abnormal CT scan or physical examination may be asked to undergo a tumor biopsy (surgical removal of a piece of tumor tissue) for research purposes.

DETAILED DESCRIPTION:
Background:

Over 80% of patients with advanced stage epithelial ovarian cancer will relapse

Serum biomarkers are needed for predictors of persistent disease and relapse

CA-125 is a less than satisfactory clinical tool for detecting relapse

A serum repository of samples from women with ovarian cancer is needed to develop and validate the multiple tests being created for ovarian cancer recurrence and screening.

Objectives:

To create a multi-institutional repository from which investigations of serum proteomic signature profiles of epithelial ovarian cancer and relapse will be developed and validated

To determine the sensitivity and specificity of the proteomic signature profiles for relapse

To compare the accuracy of proteomic evaluation and CA125 in classifying patient disease progression

To identify the temporal relationship between a rise in CA125 value versus the development of proteomic signature profiles of relapse.

To detect the impact of study participation on quality of life.

To collect epidemiological data for patients in the target population

Eligibility:

Patients in first remission from treatment of FIGO stage III/IV primary peritoneal, fallopian tube, or epithelial ovarian carcinoma as defined by normal CA125, no evidence of disease on abdominopelvic CT scan, and normal post-hysterectomy physical exam.

Entry within 12 weeks of last administration of chemotherapy.

S/P surgical debulking and completion of primary therapy with platinum/taxane-containing chemotherapy of no more than a total of 8 cycles.

Laboratory evidence of good end organ function.

Design:

Phase of Trial: Biomarker/Laboratory Analysis.

Number of patients to be enrolled: 400

Planned statistical analysis for primary endpoint: Training set to include 100 women, half of whom are in remission and half of whom have recurrent disease. Validation set will include 200 women, half of whom are in remission and half of whom have recurrent disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1<TAB>All patients in first complete response from treatment of FIGO stage III/IV primary peritoneal, fallopian tube, or epithelial ovarian carcinoma as defined by: normal CA-125, normal post-hysterectomy physical exam, no evidence of disease on abdominopelvic CT scan (or other noninvasive reassessment, e.g. MRI). PET scans are not acceptable for confirmation of complete response.

2.1.2<TAB>Pathology of the primary tumor must be confirmed by the registering center prior to protocol entry.

2.1.3<TAB>Entry within 9 weeks of completion of final cycle of chemotherapy (within 12 weeks of last administration of chemotherapy).

2.1.4<TAB>S/P surgical debulking and completion of primary therapy with platinum/taxane -containing chemotherapy of no more than 8 total cycles.

2.1.5<TAB>Patients who undergo second look laparotomy or laparoscopy and have microscopic residual disease but who elect not to have treatment will be eligible to enroll.

2.1.6<TAB>Histology slides adequate to confirm the pathology and staging must be submitted to the coordinating center within 3 months of enrollment. (If available, a sample of frozen primary tumor should also be forwarded).

2.1.7<TAB>Patients must be able and willing to provide informed consent to participate in the trial.

2.1.8<TAB>Patients must have laboratory evidence of good end organ function by criteria in Table 1 below. The upper limit of normal is based upon each registering center's laboratory normal ranges.

Laboratory based inclusion criteria:

Laboratory Test: AST(SGOT) and ALT(SGPT)

Required value: less than or equal to 2.5 times the institutional upper limit of normal creatinine

OR

Laboratory Test: Creatinine

Required value: Less than or equal to 2.0

Laboratory Test: Creatinine clearance

Required Value: Greater than or equal to 45 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.

EXCLUSION CRITERIA:

2.2.1<TAB>Patients with nonepithelial ovarian cancer, mixed epithelial/nonepithelial ovarian cancer (i.e., Mixed Malignant Mullerian Tumors), or tumors of low malignant potential. Patients with stage I or II epithelial ovarian, fallopian tube, or primary peritoneal cancer.

2.2.2<TAB>Patients may not be receiving chemotherapy (therapeutic or consolidation), maintenance, alternative therapy, or radiation therapy. No anti-cancer therapy of any kind is allowed while the patient is on-study. Replacement hormonal therapy is allowed but must be clearly indicated on the case report forms submitted. Hormonal anti-cancer therapies such as tamoxifen and raloxifene will not be permitted while on study.

2.2.3<TAB>Patients with a life expectancy of less than 6 months for any reason.

2.2.4 <TAB>Patients with a history of other invasive malignancies within the past five years prior to enrollment except for curatively treated carcinoma in situ of the cervix, ductal or lobular carcinoma in situ of the breast, concomitant stage I endometrial cancer, or basal or squamous cell skin cancers.

2.2.5 <TAB>Complementary and alternative agent use is discouraged on this study due to the possibility that the use of these agents may alter the serum protein pattern. The Institutional Principal Investigator will have discretion as to whether complementary or alternative agent usage will prevent eligibility on a case by case basis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in first remission from treatment of FIGO stage III/IV primary peritoneal, fallopian tube, or epithelial ovarian carcinoma as defined by normal CA125, no evidence of disease on abdominopelvic CT scan, and normal post-hysterectomy physical exam.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2005-12-12 (Actual)

PRIMARY OUTCOMES:
Create a multi-institutional repository from which investigations of serum proteomic signature profiles of epithelial ovarian cancer and relapse will be developed and validated | End of specimen collection
  Multi-institutional repository from which investigations of serum proteomic signature profiles of epithelial ovarian cancer and relapse will be developed and validated

CONTACTS AND LOCATIONS:
Overall Officials: Elise C Kohn, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Evanston Northwestern University Hospital, Evanston, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Dana Farber, Boston, Massachusetts
  - New York University School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington/Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Pacific Ovarian Cancer Research Consortium at FHCRC, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data are available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Patsner B, Orr JW Jr, Mann WJ Jr, Taylor PT, Partridge E, Allmen T. Does serum CA-125 level prior to second-look laparotomy for invasive ovarian adenocarcinoma predict size of residual disease? Gynecol Oncol. 1990 Sep;38(3):373-6. doi: 10.1016/0090-8258(90)90076-w. PMID 2227551
- [Background] Petricoin EF, Ardekani AM, Hitt BA, Levine PJ, Fusaro VA, Steinberg SM, Mills GB, Simone C, Fishman DA, Kohn EC, Liotta LA. Use of proteomic patterns in serum to identify ovarian cancer. Lancet. 2002 Feb 16;359(9306):572-7. doi: 10.1016/S0140-6736(02)07746-2. PMID 11867112
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0232.html